CLINICAL TRIAL: NCT04787146
Title: File Analysis of Falling Patients: Are Drugs Frequently Involved
Acronym: ADOPAC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ADOPAC
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Fall Patients
Keywords: Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: From Monday to Friday, the study will be offered to patients selected consecutively and who have fallen within the previous 24 hours (between 7.55 a.m. the day before and 7.55 a.m. the next day).
  After delivery of the written information note to the patient, the investigating physician answers the patient's questions and accepts his non-objection. The patient should be given sufficient time to think things through to make the decision to participate in the study.
  Its non-opposition will be traced in the computerized medical file created on the day of its inclusion in the protocol. Each patient participating in the study retains the possibility of participating simultaneously in another research. No exclusion period is provided for in the protocol.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Once the patient is included, a drug assessment is carried out as part of the treatment and then an compliance questionnaire is submitted to him.

SUMMARY:
The damage caused by patient falls is a major public health problem, due to the large and growing number of people concerned, the potentially serious consequences but also the financial cost generated by their care.

These consequences can be physical as well as psychological. Fractures and pain are the first consequences that come to mind, but many others should be mentioned: post-fall syndrome, loss of autonomy or even entering an institution, fear of falling, loss of confidence in itself.

DETAILED DESCRIPTION:
During 2018, 285 reports of falls were counted within the Paris Saint-Joseph Hospital Group (GhPSJ). Reducing these falls is one of the institutional goals. A dedicated working group has been created to put in place preventive and corrective measures.

These falls can be caused by many factors to the patient:

1. Intrinsic:

   * History of a fall,
   * pathologies (Parkinson's or Alzheimer's disease),
   * hearing and visual disturbances,
   * urinary incontinence.
2. extrinsic:

   * Unsuitable shoes
   * unsuitable habitat,
   * slippery floors (eg bathroom).

Among the intrinsic factors, polypharmacy is also found. It has been established that certain drug classes are at risk of falling, in particular psychotropic drugs (benzodiazepines, hypnotics, anxiolytics, antidepressants, neuroleptics) which promote sedation and dizziness, hypoglycemic drugs which cause hypoglycaemia in diabetic patients on -treated or antihypertensive drugs causing hypotension.

It is now clearly established that drug adherence to treatment is poor in cities, giving rise to omissions but also sometimes to overconsumption of certain drugs, including psychotropic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* French-speaking patient
* Patient hospitalized within the Paris Saint-Joseph Hospital Group
* Patient who fell during hospitalization and for whom a fall report has been completed

Exclusion Criteria:

* Patients in the process of therapeutic limitation
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient objecting to participation in the study
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From Monday to Friday, the study will be offered to patients selected consecutively and who have fallen within the previous 24 hours (between 7.55 a.m. the day before and 7.55 a.m. the next day).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
To assess the prevalence of falls associated with one or more risk factors for drug iatrogenism within the Paris Saint-Joseph Hospital Group. | 1 week
  Percentage of falls involving one or more drugs at risk of falling

SECONDARY OUTCOMES:
List the drug treatments at risk taken by patients who fall | 1 week
  To list the drug treatments taken by the patients who fall: carrying out the patient's drug assessment
Evaluate the relevance of drug prescriptions in patients who fall | 1 week
  Average number of inappropriate medication prescriptions per patient
Evaluate the overall compliance of falling patients | 1 week
  Average compliance score in patients who fall

CONTACTS AND LOCATIONS:
Overall Officials: Elodie MENAGE, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France